CLINICAL TRIAL: NCT06220123
Title: A Multicenter, Randomized, Open-label, Active-controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of SHR-2004 Injection in Preventing Postoperative Venous Thromboembolism in Patients Undergoing Ovarian Cancer Surgery
Brief Title: A Study to Evaluate the Efficacy and Safety of SHR-2004 Injection in Preventing Postoperative Venous Thromboembolism in Patients Undergoing Ovarian Cancer Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Suncadia Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SHR-2004-202
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Preventing Postoperative Venous Thromboembolism in Patients Undergoing Ovarian Cancer Surgery
MeSH Terms: interventions — enoxaparin sodium; Rivaroxaban

STUDY DESIGN:
Intervention Model Description: 1:1 randomized and paralleled 2 arms: Investigational product arm， Positive control arm
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational product arm (Experimental)
  Interventions: Drug: SHR-2004
- Positive control arm (Active Comparator)
  Interventions: Drug: Enoxaparin Sodium Injection; Rivaroxaban Tablets

INTERVENTIONS:
Drug: SHR-2004 — Investigational product arm: SHR-2004
  Arms: Investigational product arm
Drug: Enoxaparin Sodium Injection; Rivaroxaban Tablets — Positive control arm: Enoxaparin Sodium Injection + Rivaroxaban Tablets
  Arms: Positive control arm

SUMMARY:
This study is designed to evaluate the efficacy and safety of SHR-2004 injection in preventing postoperative venous thromboembolism in patients undergoing ovarian cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years old on the day of signing the informed consent form;
2. Diagnosed as stage III-IV or recurrent ovarian cancer;
3. Have surgical indications and no contraindications to surgery, and voluntarily undergo laparotomy or laparoscopic surgery to treat ovarian cancer;
4. Understand the research procedures and methods, voluntarily participate in this trial, and sign the written informed consent form.

Exclusion Criteria:

1. The primary site of the tumor is not the ovary or there is brain metastasis;
2. A history that may increase the risk of bleeding;
3. A history of VTE in the past or during screening, or a disease that increases thrombosis tendency such as protein C deficiency;
4. Patients with atrial fibrillation requiring anticoagulant treatment or the use of artificial heart valves during screening;
5. Acute coronary syndrome within 3 months;
6. Poorly controlled hypertension before screening, and uncontrolled hypertension within 6 months severe cardiac arrhythmia;
7. Any laboratory test indicator during screening or baseline does not meet the standards in the exclusion criteria;
8. Have had a history of adverse reactions or allergies related to rivaroxaban or enoxaparin, such as heparin-induced thrombocytopenia;
9. Have used any drugs prohibited other than investigational drugs within 7 days before screening or plan to use during the study;
10. Those who have participated in any drug intervention clinical trial within 1 month before screening, or those who are within 5 half-lives of the investigational drug at the time of screening, Whichever is longer;
11. Those who are expected to use postoperative neuraxial analgesia;
12. Those who are expected to use plantar vein pumps, intermittent pneumatic compression devices, electronic or mechanical muscle stimulators after surgery;
13. Other circumstances in which the researcher believes that the subject is not suitable to participate in this trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Primary efficacy endpoint: The incidence rate of VTE from the first medication to the end of the treatment period (Day 28) | up to Day 28
  including asymptomatic deep vein thrombosis (DVT) (confirmed by bilateral lower limb venous compression ultrasound), objectively confirmed symptomatic DVT, and objectively confirmed non-fatal. The composite endpoint of pulmonary thromboembolism (PE) and VTE-related death.
The composite endpoint incidence rate of major bleeding and clinically relevant non-major bleeding events as defined by the International Society on Thrombosis and Haemostasis (ISTH) from the first dose to the end of the treatment period | up to Day 28
  Primary safety endpoints

SECONDARY OUTCOMES:
The event rate of each component of the primary efficacy endpoint | up to Day 28
  Secondary efficacy endpoint
Secondary efficacy endpoint: The total VTE incidence rate from the first medication to the end of follow-up (D85) and the incidence rate of each component event | up to Day 85
  including asymptomatic DVT (confirmed by bilateral lower limb venous compression color ultrasound), objectively confirmed symptomatic DVT, and objectively confirmed non-fatal. The composite endpoint of sexual PE and VTE-related death.
The event rate of each component of the primary safety endpoint | up to Day 28
  Secondary safety endpoints
The incidence of any bleeding events (including minor bleeding events) from the first dose to the end of the treatment period | up to Day 28
  Secondary safety endpoints
The composite endpoint incidence rate and each component event rate of major bleeding and clinically relevant non-major bleeding events that meet the definition of ISTH from the first medication to the end of follow-up | up to Day 85
  Secondary safety endpoints
The incidence of any bleeding events (including minor bleeding events) from the first dose to the end of follow-up | up to Day 85
  Secondary safety endpoints
The incidence and severity of adverse events. | up to Day 85
  Secondary safety endpoints

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided